CLINICAL TRIAL: NCT03164876
Title: A Randomised, Double-blind, Placebo-controlled Study of the Safety, Pharmacokinetics and Exploratory Pharmacodynamics of AUT00206 for 28 Days as Adjunctive Therapy in Patients With Recently Diagnosed Schizophrenia
Brief Title: Safety, Tolerability and Pharmacokinetics of AUT00206 in Patients With Schizophrenia, and Also Explores the Effects of AUT00206 on Relevant Central Biomarkers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUT031206
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose AUT00206 800 mg BD (Experimental): AUT00206 800mg twice daily for 28 days
  Interventions: Drug: AUT00206
- Placebo (Placebo Comparator): Placebo to match AUT00206 twice daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUT00206 — 4 capsules of 200mg AUT00206, twice daily, to take orally with food for 4 weeks
  Arms: Dose AUT00206 800 mg BD
Drug: Placebo — 4 capsules of placebo, twice daily, to take orally with food for 4 weeks
  Arms: Placebo

SUMMARY:
This study will investigate the safety, tolerability, PK and PD profile of AUT00206 after repeated doses in patients with stable but symptomatic schizophrenia, taking one or two established anti-psychotic drugs. The subjects will undergo brain imaging, tests of cognition and tests of auditory function and electrophysiological measures in addition to routine safety monitoring. Because of the pioneering and novel mechanism of action of this drug, a key objective is to characterize this range of biomarkers which will inform the future development of the drug.

ELIGIBILITY:
Key inclusion Criteria:

* Male patients with a diagnosis of schizophrenia no more than 5 calendar years (before screening);
* Positive and negative symptoms assessed by PANSS;
* Medically and psychiatrically stable;
* On a stable dose of antipsychotic drugs;
* Able to give fully informed written consent and likely to comply with the requirements of the trial.

Key exclusion Criteria:

* clinically relevant, as assessed by a physician, abnormal findings at the screening assessment;
* sensitivity to excipients of the trial medication;
* current use of contraindicated drugs;
* participation in another clinical trial of unlicensed medicines within the previous 30 days;
* loss of more than 400 mL blood, within the previous 3 months; history of drug or alcohol dependence in the last year;
* significant acute or chronic illness;
* significant medical history or concurrent medical condition that warrants exclusion;
* objection by subject's physician

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male 18-50 Years
Enrollment: 24 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events over 28 days treatment of AUT00206 compared to Placebo | 28 days
Plasma concentrations of AUT00206 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London Institute of Psychiatry, Psychology and Neuroscience (IoPPN), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No